CLINICAL TRIAL: NCT05528523
Title: The Relationship Competences Guiding Tool: A Development, Content Validation and Implementation Study
Brief Title: The Relationship Competences Guiding Tool
Acronym: NarratUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Ana Choperena, Principal investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020.002
Record Dates: First submitted 2022-08-24; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Nurse-Patient Relations; Professional Role; Narration
Keywords: Patient centred care; Clinical narrative; Guide
MeSH Terms: conditions — Narration

STUDY DESIGN:
Masking Description: Researchers were avoided to have all data in order not to prejudge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Writing a clinical narrative (Other): The participants had to write a clinical narrative regarding a significant encounter with a patient.
  Interventions: Other: Writing a clinical narrative

INTERVENTIONS:
Other: Writing a clinical narrative — The participants had to write a clinical narrative regarding a significant encounter with a patient.

SUMMARY:
Aim: The aims of this study are: (1) to present the development, content validation and implementation study of the Relationship Competences Guiding Tool (RCGT); (2) to show some examples of how each of the items of the guide may be reflected on clinical narratives written by nurses, and justify its corresponding scores after the evaluation; (3) to present how the language and content of the narratives are interpreted with this guide and to describe an exemplar; (4) to present barriers and facilitators of its application.

Background: From a person-centred care approach, the fostering of authentic relationships with patients is key for therapeutic benefits. Therefore, it is essential to help nurses to establish meaningful relationships with patients and help them to achieve these abilities. In this line, clinical narratives can be used as a way to promote reflective practice and professional competences development between nurses. A guide to evaluate the knowledge, skills, attitudes and values necessary for developing authentic encounters with patients reflected by nurses on clinical narratives was developed and implemented.

Design: Design and evaluation of the RCGT, and evaluation of its implementation Methods: This study was conducted in three major steps. Step one entailed the conceptualization. Step two included the generation of items and content validation. Then, in step three, the tool was used to independently evaluate 25 narratives by two researchers, in order to identify and exemplify the attributes of the nurse patient relationship defined on the guide and identify barriers and facilitators. One of the narratives was linguistically analysed in the light of the guide, in order to provide a comprehensive view of the interpretative strategies deployed by evaluators.

Results: The RCGT helped to identify nursing professional competences reflected in clinical narratives. The tool guided in the process of assigning scores to the corresponding items. The use of the tool helped to identify some barriers and facilitators before and during the narrative evaluation process.

Conclusions: A clear, relevant, conceptually and linguistically adequate guide for assessing clinical narratives was obtained. The RCGT can be applied to accurately interpret how nurses reflect professional competences in a clinical narrative as a preliminary step to design a measurement tool.

DETAILED DESCRIPTION:
This study is the first to present a valid guide for interpreting the essential aspects (respect, intentional presence and knowing the person) of the nurse-person relationship using clinical narratives. This is therefore an innovative tool to facilitate the nurses' work in caring patients and families, ensuring the success of a person-centred care for the target population. Moreover, this study describes the rigorous process that has been carried out both for the content validation of the RCGT, as well as for its application by two researchers independently with different backgrounds and perspectives.

ELIGIBILITY:
Inclusion Criteria:

* nurses who agreed to participate and signed informed consent.
* nurses from different hospitals and clinical departments/services, such as general hospital wards, intensive care units, outpatient services, and other departments (i.e., perioperative, elder care, and haemodialysis, emergency, etc).

Exclusion Criteria:

. other health professionals different from nurses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Professional competence 1: respect | One month
  The knowledge, skills, attitudes and values necessary for developing respect towards the patient. The Relationship Competences Guiding Tool was used to evaluate this competence.

OTHER OUTCOMES:
Professional competence 2: intentional presence | One month
  The knowledge, skills, attitudes and values necessary for developing intentional presence towards the patient. The Relationship Competences Guiding Tool was used to evaluate this competence.
Professional competence 3: knowing the person | One month
  The knowledge, skills, attitudes and values necessary for knowing the person. The Relationship Competences Guiding Tool was used to evaluate this competence.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Choperena, PhD, Principal Investigator — University of Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
We will not share the clinical narratives. We will use the conclusions of the study for educational purposes.

REFERENCES:
- [Background] Choperena A, Oroviogoicoechea C, Zaragoza Salcedo A, Olza Moreno I, Jones D. Nursing narratives and reflective practice: A theoretical review. J Adv Nurs. 2019 Aug;75(8):1637-1647. doi: 10.1111/jan.13955. Epub 2019 Feb 27. PMID 30666703
- [Background] Choperena A, Pardavila-Belio MI, Errasti-Ibarrondo B, Oroviogoicoechea C, Zaragoza-Salcedo A, Goni-Viguria R, Martin-Perez S, Llacer T, La Rosa-Salas V. Implementation and evaluation of a training programme to promote the development of professional competences in nursing: A pilot study. Nurse Educ Today. 2020 Apr;87:104360. doi: 10.1016/j.nedt.2020.104360. Epub 2020 Jan 29. PMID 32135456